CLINICAL TRIAL: NCT07219849
Title: A Two-part Adaptive Double-blind Randomized Placebo-controlled Study to Assess the Appropriate Dose and the Appropriate Dosing Frequency of ALDP 001 in Adults With Seasonal Allergic Rhinitis (SAR) Assessed Using an Allergen Challenge Chamber/EEC
Brief Title: A Study to Determine the Optimal Dose and Frequency of ALDP001 Nasal Spray in Adults With Seasonal Allergic Rhinitis Under Allergen Exposure
Acronym: ALDP001
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alixer Nexgen Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK45-ALDP001/ C2D05456
Record Dates: First submitted 2025-10-17; First posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Seasonal Allergic Rhinitis (SAR)
Keywords: ALDP001 Nasal Spray
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind pharmacy controlled randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ALDP001 0.125% w/v (Experimental): Participants will self-administer one spray in each nostril, either once or twice daily, using the assigned nasal spray kit for a duration of eight days
  Interventions: Drug: ALDP001 Nasal Spray
- ALDP001 (0.25% w/v) (Experimental): Participants will self-administer one spray in each nostril, either once or twice daily, using the assigned nasal spray kit for a duration of eight days
  Interventions: Drug: ALDP001 Nasal Spray
- ALDP001 (0.5% w/v) Nasal Spray (Experimental): Participants will self-administer one spray in each nostril, either once or twice daily, using the assigned nasal spray kit for a duration of eight days
  Interventions: Drug: ALDP001 Nasal Spray
- Placebo Nasal Spray (Placebo Comparator): Participants will self-administer one spray in each nostril, either once or twice daily, using the assigned nasal spray kit for a duration of eight days
  Interventions: Drug: Placebo Nasal spray

INTERVENTIONS:
Drug: ALDP001 Nasal Spray — Experimental Arm
  Arms: ALDP001 (0.25% w/v); ALDP001 (0.5% w/v) Nasal Spray; ALDP001 0.125% w/v
Drug: Placebo Nasal spray — Controlled arm
  Arms: Placebo Nasal Spray

SUMMARY:
This study aims to evaluate the effectiveness and safety of ALDP001 Nasal Spray in treating seasonal allergic rhinitis, and to identify the optimal dosage and administration frequency for this formulation.

DETAILED DESCRIPTION:
The study will be conducted in two Parts. In Part A, participants will receive a once-daily (OD) dose of the nasal spray for eight days. An interim analysis will then be performed to identify the optimal dose for the next part. In Part B, participants will be administered a twice-daily (BD) dose of the selected formulation from Part A to evaluate the appropriate dosing frequency for the regimen.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Allergic Rhinitis (AR), as determined by the presence of seasonal rhinitis symptoms for several months per year, for more than 1 year and are not attributed to infections or nasal abnormalities
* Positive skin prick test (SPT) response to ragweed pollen (allergen induced wheal diameter at least 3 mm larger than the negative control) in the previous 12 months
* Healthy as determined by a responsible and experienced Investigator, based on a medical evaluation including medical history, physical examination, vital signs, ECG, and lab tests.

Exclusion Criteria:

* Nasal abnormalities likely to affect the outcome of the study, i.e. nasal septal perforation, nasal polyps, sinusitis and other nasal malformations.
* History of frequent nosebleeds.
* Participants with rhinitis medicamentosa.
* Current or chronic history of hepatic disease.
* A QTcF (Fridericia-corrected QT interval) >450 ms in males or >470 ms in females.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Total Nasal Symptom Score | Day 9
  Total Nasal Symptom Score (TNSS) is calculated by summing scores from four nasal symptoms: itchy nose, nasal congestion, runny nose, and sneezing. Each symptom is rated on a scale from 0 to 3, where:
  0 - None (no symptoms)
  1. - Mild (minimal awareness, easily tolerated)
  2. - Moderate (noticeable and bothersome, but tolerable)
  3. - Severe (difficult to tolerate, interferes with daily activities or sleep)
  The total score ranges from 0 to 12. Participants will record TNSS at multiple timepoints: 0, 30, 60, 90, 120, 180, and 240 minutes, both at baseline and after 8 days of treatment.
  The change from baseline (CFB) at each timepoint will be calculated and compared between study arms to evaluate the treatment effect of ALDP001 Nasal Spray.

SECONDARY OUTCOMES:
Change from baseline in the Area Under the Curve of the Total Nasal Symptom Score at Day 9 | Day 9
  The Area Under the Curve (AUC) for the Total Nasal Symptom Score (TNSS) will be calculated based on measurements taken at multiple timepoints: 0, 30, 60, 90, 120, 180, and 240 minutes, both at baseline and after 8 days of treatment. The TNSS is a composite score assessing nasal symptoms including congestion, rhinorrhea, itching, and sneezing. Each symptom is rated on a scale from 0 (no symptoms) to 3 (severe symptoms), resulting in a total score range of 0 to 12, where higher scores indicate worse nasal symptoms. The change from baseline in the AUC for TNSS after the treatment period will be analyzed and compared across study arms to assess the efficacy of the intervention. A lower AUC value indicates better symptom control, and the AUC is expected to be lowest for the optimum dose group, reflecting improved treatment efficacy. The change from baseline in AUC of the TNSS for each dose group will be analyzed to identify the optimum dose.

OTHER OUTCOMES:
Number of participants with Adverse events (AEs), with abnormal Clinical Laboratory Parameters, abnormal ECG readings | From enrollment to End of Study i.e. 10 days
  The number of participants who experience adverse events (AEs), as well as those presenting with abnormal clinical laboratory parameters (including hematology, biochemistry, and urinalysis) and abnormal ECG findings (such as QT interval prolongation), will be recorded and analyzed to evaluate the safety profile of the investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Couroux, MD, Principal Investigator — Cliantha Research
Locations (1):
- Cliantha Research, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
masked Lab reports, masked Total Nasal symptom Score etc